CLINICAL TRIAL: NCT04975009
Title: Localizing and Modulating Competing Memories of Fear and Safety in the Human Brain
Brief Title: Neuroimaging Memories of Fear and Safety in the Human Brain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Texas at Austin (Other)
Responsible Party: Principal Investigator, Joseph E. Dunsmoor, Jr., Assistant Professor of Psychiatry, University of Texas at Austin
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2020020157-MODCR01
Record Dates: First submitted 2021-07-06; First posted 2021-07-23 (Actual); Last update posted 2022-05-17 (Actual); Status verified 2022-05

CONDITIONS: Fear Anxiety; PTSD
Keywords: Pavlovian conditioning; Fear Conditioning; Neuroimaging
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PTSD group (Experimental): Participants will be screened and diagnosed using typical screening procedures and diagnostic criteria (e.g., the clinically administered PTSD scale). Participants also screened for contraindications for MRI. The learning paradigm inside the MRI scanner occurs over 3 days. The first two days are consecutive (back-to-back) and the third MRI visit is 1 month later. Participants are asked to look at a screen and listen to simple tones over headphones, while the experimenter measures brain activity and physiological measures of arousal (e.g., sweating from sensors on the hand). These visits will be scheduled within two weeks from the baseline and assessment visit.
  Interventions: Behavioral: Fear conditioning
- Healthy control group (Experimental): Participants will be healthy adults without a history of psychiatric illness. Participants also screened for contraindications for MRI. The learning paradigm inside the MRI scanner occurs over 3 days. The first two days are consecutive (back-to-back) and the third MRI visit is 1 month later. Participants are asked to look at a screen and listen to simple tones over headphones, while the experimenter measures brain activity and physiological measures of arousal (e.g., sweating from sensors on the hand). These visits will be scheduled within two weeks from the baseline and assessment visit.
  Interventions: Behavioral: Fear conditioning

INTERVENTIONS:
Behavioral: Fear conditioning — Participants will learn to associate neutral stimuli with a mildly uncomfortable electrical stimulation to the wrist. The intensity of the electrical stimulus is calibrated prior to the start of the experiment to a level deemed highly annoying but not painful by the participant.

SUMMARY:
The purpose of this research is to use functional magnetic resonance imaging (fMRI) to investigate how the brain forms associations between neutral and negative stimuli. The ultimate goal is to understand the neural systems involved in regulating negative emotional responses to fearful stimuli.

DETAILED DESCRIPTION:
This study uses functional magnetic resonance imaging (fMRI) to investigate how the brain forms associations between neutral stimuli and a mildly uncomfortable electrical stimulation to the wrist. Referred to as Pavlovian fear conditioning. The goal is to compare brain activity between individuals with posttraumatic stress disorder (PTSD) and healthy control subjects without PTSD. PTSD is characterized by excessive fear and anxiety, including in harmless situations. The data here will help us better understand dysregulation in neural circuitry involved in fear recovery, which has implications for improving treatment.

ELIGIBILITY:
Inclusion Criteria (All study populations):

1. Volunteers with a major medical illness or a neurological disorder (e.g., Parkinson's Disease), or neurological abnormality including significant head trauma (loss of consciousness > 5 min).
2. A positive pregnancy test in female volunteers.
3. Benzodiazepines, tested using urine tox screen.
4. For the healthy subjects, exclusion is meeting criteria for either PTSD, or any other psychiatric disorder, or any prior psychiatric hospitalizations.
5. For the healthy subjects, exclusion is prior use of a psychotropic medication for longer than 1 month.
6. History of moderate to severe cannabis use disorder.
7. Magnetic Resonance Imaging (MRI) exclusions: Claustrophobia; tattoos above the shoulders; permanent eyeliner or permanent; artificial eyebrows; cardiac pacemaker; metal fragments in eye, skin, or body, including shrapnel; heart valve replacement; brain clips; venous umbrella; being a sheet-metal worker or welder; lifetime history of aneurysm surgery; intracranial bypass, renal, or aortic clips; prosthetic devices such as middle ear, eye, joint, or penile implants; joint replacements; non-removable hearing aid, neurostimulator, or insulin pump; shunts/stents; metal mesh/coil implants; metal plate/pin/screws/wires; or any other metal implants.

Inclusion Criteria (PTSD populations):

1. Meet diagnostic criteria for PTSD, as assessed by standard diagnostic instruments.
2. Participants with PTSD are eligible if they meet diagnostic criteria for current PTSD. This is determined by the presence of a Criterion A event in addition to a severity score of 2 or greater on 1 symptom in clusters B and C and on 2 symptoms in clusters D and E, in addition to meeting criteria F and G. The specific form of trauma is not considered for inclusion/exclusion.
3. Volunteers in the patient group, but not healthy control group, may also meet criteria for a mood disorder (except for bipolar affective disorder, see exclusions below), as well as other anxiety disorders (panic disorder, agoraphobia, social phobia, generalized anxiety disorder, or obsessive compulsive disorder). Including these comorbidities is essential because of the high frequency of co-occurring mood and anxiety disorders with PTSD.

Exclusion Criteria (all participants):

1. Volunteers with a major medical illness or a neurological disorder (e.g., Parkinson's Disease), or neurological abnormality including significant head trauma (loss of consciousness > 5 min).
2. A positive pregnancy test in female volunteers.
3. Benzodiazepines, tested using urine tox screen.
4. For the healthy subjects, exclusion is meeting criteria for either PTSD, or any other psychiatric disorder, or any prior psychiatric hospitalizations.
5. For the healthy subjects, exclusion is prior use of a psychotropic medication for longer than 1 month.
6. History of moderate to severe cannabis use disorder.
7. MRI exclusions: Claustrophobia; tattoos above the shoulders; permanent eyeliner or permanent; artificial eyebrows; cardiac pacemaker; metal fragments in eye, skin, or body, including shrapnel; heart valve replacement; brain clips; venous umbrella; being a sheet-metal worker or welder; lifetime history of aneurysm surgery; intracranial bypass, renal, or aortic clips; prosthetic devices such as middle ear, eye, joint, or penile implants; joint replacements; non-removable hearing aid, neurostimulator, or insulin pump; shunts/stents; metal mesh/coil implants; metal plate/pin/screws/wires; or any other metal implants.

Exclusion Criteria (PTSD group):

* 1. Volunteers meeting DSM-5 criteria for history of or current psychotic or bipolar affective disorders, a current eating disorder (bulimia, anorexia nervosa), or dissociative identity disorder.

  2. Volunteers meeting DSM-5 criteria for another substance use disorder, with the exception of caffeine or nicotine, within the past 12 months.

  3. Individuals considered an immediate suicide risk based on the Columbia Suicide Severity Scale (C-SSRS) or who would likely require hospitalization during the course of the study.

  4. Participants must be stable on medication.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 240 (Estimated)
Dates: Start 2021-07-12 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in physiological arousal throughout the experimental phases, compared between healthy controls and PTSD participants | through study completion, an average of 1 month.
  Skin conductance responses measure sweating throughout the experiment. We compare the magnitude of this response during each phase of the experiment between groups.
Change in functional MRI data in fear-learning circuitry throughout the experimental phases, compared between healthy controls and PTSD participants | through study completion, an average of 1 month.
  Participants undergo scanning on a 3-Tesla MRI during all experimental phases. Blood-oxygen-level-dependent (BOLD) signal in key brain regions will be compared between groups.

SECONDARY OUTCOMES:
Individual differences in brain-behavior responses | through study completion, an average of 1 month.
  Individual participants arousal, as well as trait variable of anxiety and symptom severity, will be used as a covariate in neuroimaging analyses to assess brain-behavior correlations.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - The University of Texas at Austin, Austin, Texas
  - Biomedical Imaging Center, Austin, Texas